CLINICAL TRIAL: NCT07066644
Title: Intraoperative Pathologic Evaluation of Central Lymph Nodes to Determine the Extent of Surgery in Papillary Thyroid Carcinoma : A Retrospective Cohort Study
Brief Title: Intraoperative Pathologic Evaluation of Central Lymph Nodes in Papillary Thyroid Carcinoma
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Kyu Eun Lee, Professor, Seoul National University Hospital
Other Study IDs: H-2309-109-1467
Record Dates: First submitted 2025-06-23; First posted 2025-07-15 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Thyroid Cancer, Papillary
Keywords: central lymph node metastasis; intraoperative pathological evaluation
MeSH Terms: conditions — Thyroid Cancer, Papillary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: central node dissection — dissection of level VI compartment by AAHNS (American association of head and neck surgeons) classification

SUMMARY:
Efficacy of Intraoperative pathologic evaluation of central lymph nodes

DETAILED DESCRIPTION:
This study aimed to evaluate the effectiveness of intraoperative pathological examination and determine the risk factors for central lymph node metastasis in patients with unilateral clinically node-negative (cN0) papillary thyroid carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* patients with unilateral papillary thyroid cancer
* no evidence of lymph node metastasis (clinically N0)
* performed with Intraoperative pathologic evaluation

Exclusion Criteria:

* those with a history of neck surgery
* those with lateral lymph node metastasis
* those with suspected extrathyroidal extension
* those in whom Intraoperative pathologic evaluation was not performed

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: the patients with unilateral papillary thyroid cancer classified as cN0 and performed with Intraoperative pathologic evaluation
Sampling Method: Probability Sample
Enrollment: 509 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
the accuracy of IOPE | Perioperative
  To evaluate IOPE accuracy, the findings were compared with the final pathology results, utilizing key parameters such as sensitivity, specificity, false-negative rate (FNR), and false-positive rate for analysis.

SECONDARY OUTCOMES:
the incidence of complications in IOPE [safety of IOPE] | up to 6 months
  The safety was evaluated by examining the incidence of complications, including vocal cord palsy and hypoparathyroidism.
  vocal cord palsy : measured by laryngeal sono hypoparathyroidism : serum parathyroid hormone levels < 15.0 pg/mL
the risk factors for central lymph node metastasis | perioperative
  To determine the risk factors for central lymph node metastasis, univariate and multivariate logistic regression analyses were performed to identify the correlations between clinicopathological characteristics and the final pathological presence of central lymph node metastasis.
  clinicopathological factors : sex, age (<55, ≥55), sonographic features, size (<1cm, ≥1cm) presence of central lymph node metastasis was confirmed by final pathology

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Jongno-gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ahn BH, Kim JR, Jeong HC, Lee JS, Chang ES, Kim YH. Predictive factors of central lymph node metastasis in papillary thyroid carcinoma. Ann Surg Treat Res. 2015 Feb;88(2):63-8. doi: 10.4174/astr.2015.88.2.63. Epub 2015 Jan 27. PMID 25692116
- [Result] Bae HL, Ahn JH, Kwak J, Kim HS, Yoon SG, Yi JW, Kim SJ, Lee KE. Intraoperative pathologic evaluation of central compartment lymph nodes in patients undergoing lobectomy for unilateral papillary thyroid carcinoma. Asian J Surg. 2024 Jan;47(1):360-366. doi: 10.1016/j.asjsur.2023.08.203. Epub 2023 Oct 25. PMID 37891110